CLINICAL TRIAL: NCT03869528
Title: A Randomized Controlled Trial to Evaluate the Efficacy of Topical Pharyngeal Anaesthesia Using 5 vs 10 Sprays of 10% Lignocaine During Flexible Bronchoscopy
Brief Title: 5 Versus 10 Sprays of Lignocaine for Pharyngeal Anaesthesia During Bronchoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Karan Madan, Dr Karan Madan, Assistant Professor, Department of Pulmonary Medicine and Sleep Disorders, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 510 RCT
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Bronchoscopy; Anesthesia, Local
Keywords: bronchoscopy; lignocaine
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Group allocation by opaque sealed envelopes. Participant and bronchoscopist shall be unaware of the number of sprays administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5 sprays (Active Comparator): 5 sprays of 10% lignocaine administered for topical anaesthesia during flexible bronchoscopy
  Interventions: Drug: 5 sprays of 10% lignocaine
- 10 sprays (Experimental): 10 sprays of 10% lignocaine administered for topical anaesthesia during flexible bronchoscopy
  Interventions: Drug: 10 sprays of 10% lignocaine

INTERVENTIONS:
Drug: 5 sprays of 10% lignocaine — 5 sprays of 10% lignocaine
  Other Names: 5 sprays
  Arms: 5 sprays
Drug: 10 sprays of 10% lignocaine — 10 sprays of 10% lignocaine
  Other Names: 10 sprays
  Arms: 10 sprays

SUMMARY:
Flexible bronchoscopy is one of the most widely performed procedures for diagnosis of various bronchopulmonary diseases. Most patients tolerate the procedure well although cough is often reported as a distressing symptom. It is likely that the acceptance of bronchoscopy would be significantly improved with control of cough.

Topical lignocaine is administered during bronchoscopy for local anaesthesia. There is uncertainty regarding the adequate dose of lignocaine sprays for pharyngeal anaesthesia during flexible bronchoscopy. This study would help to determine the optimal dose of lignocaine sprays for pharyngeal anaesthesia during flexible bronchoscopy.

DETAILED DESCRIPTION:
For all patients meeting the inclusion criteria, the demographic profile including age, sex, weight and the type of procedures performed during bronchoscopy shall be recorded. A written informed consent will be obtained from all participants. Enrolled patients will be randomized to receive either 5 or 10 sprays of 10% lignocaine to the pharynx. This will be followed by the standard topical anesthesia procedure followed in our institution involving 5ml of 2% lignocaine gel into the nostril. Transnasal flexible bronchoscopy will be performed with additional 1% lignocaine administered as "spray as you go" method. This will be given as 2 ml aliquots- with similar volume in both groups as baseline. Procedure shall be performed with administration of sedation using Midazolam and Fentanyl if required. Primary outcome will be assessed by noting the operator rated overall procedure satisfaction as a VAS scale score.

ELIGIBILITY:
Inclusion Criteria:

* All adults ≥ 18 yrs of age undergoing flexible bronchoscopy

Exclusion Criteria:

* Uncontrolled hypertension Systolic Blood Pressure >180 mm Hg
* Symptomatic coronary artery disease
* Pregnancy
* Not giving informed consent for the procedure
* Hypoxemia (oxygen saturation [by pulse oximetry] < 92% with Fio2 of ≥ 0.3
* Bronchoscopy performed through an artificial airway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Operator rated overall procedure satisfaction | At study completion at approximately 4 months
  Visual Analogue Scale score (VAS) between 0 to 100

SECONDARY OUTCOMES:
Operator rated cough | At study completion at approximately 4 months
  Visual Analogue score (VAS) between 0 to 100
Time from bronchoscope introduction to reaching the vocal cords | At study completion at approximately 4 months
  Time in seconds
Patient willingness to return for repeat bronchoscopy | At study completion at approximately 4 months
  Proportion of patients willing for repeat bronchoscopy in each group
Cumulative lignocaine dose | At study completion at approximately 4 months
  Total dose of lignocaine in milligram (mg)
Complications | At study completion at approximately 4 months
  Proportion of patients with complications in each group

CONTACTS AND LOCATIONS:
Overall Officials: Randeep Guleria, MD DM, Study Chair — AIIMS, New Delhi
Locations (2):
- India (2):
  - AIIMS, New Delhi
  - AIIMS Rishikesh, Rishikesh

IPD SHARING:
Plan to Share IPD: No